CLINICAL TRIAL: NCT01992003
Title: Assessing the Accuracy of the Butterfly Sensor With RevK Version for Non-Invasive Hemoglobin Monitoring
Brief Title: Butterfly Sensor With Rev K Version
Status: Terminated | Type: Observational
Why Stopped: Interim analysis indicated accuracy unchanged from previous versions
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00524F
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing spine surgery

SUMMARY:
The primary purpose of this study is to assess the accuracy of the newly released Masimo SpHb Butterfly Sensor with RevK version and compare the results to a blood hemoglobin level analyzed in the UCSF Clinical Laboratories. A secondary purpose is to assess the blood hemoglobin using the Masimo Pronto-7 hand-held device immediately prior to surgery.

DETAILED DESCRIPTION:
* Masimo SpHb™ continuous hemoglobin monitoring The Masimo SpHb™ monitor with the Butterfly Sensor with RevK version will be used to continuously monitor hemoglobin electronically. The Butterfly Sensor will be connected to the 3rd or 4th finger on either the right or left hand.
* Masimo Pronto-7™ intermittent hemoglobin monitoring The Masimo Pronto-7™ is a hand-held, noninvasive device used for intermittent measuring of blood hemoglobin. The device is connected to a re-usable sensor which is clipped onto a finger for quick spot-check readings. A reading from the Pronto-7 will be taken immediately before surgery.
* Blood sampling for hemoglobin determination For the study, about a ½ tsp of blood will be collected from the arterial line placed for the purpose of surgery approximately every hour during the surgery to obtain a hemoglobin measurement to be analyzed in the UCSF Clinical Lab.

ELIGIBILITY:
Inclusion Criteria:

* Male of non-pregnant female 18 y/o or older
* American Society of Anesthesiologists Classification 1,2 or 3
* Scheduled to undergo spine or hip surgery

Exclusion Criteria:

* Pregnant or nursing
* Patients who in the investigators clinical judgement would not be suitable for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this study is to assess the accuracy of the newly released Masimo SpHb Butterfly Sensor with RevK version and compare the results to a blood hemoglobin level. | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States